CLINICAL TRIAL: NCT02545348
Title: Evaluation (Good Medical Practice Evaluation) of the Use of the Sentinel Node Biopsy in Early Stage Endometrial Cancer and Its Implication on the Adjuvant Treatement and on the Outcomes of the Cancer
Brief Title: Use of the Sentinel Node Biopsy for Early Endometrial Cancer.
Acronym: SNE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Luyckx, Assistant Chief Resident - Gynecologic Oncology - King Albert Institute, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Other Study IDs: StLucGsendo1
Record Dates: First submitted 2015-09-03; First posted 2015-09-09 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Cancer of Endometrium
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Sentinel Lymph Node Biopsy — First, the detection of the sentinel node will be preformed at the beginning of the surgery. Differents detection methods are use and the efficacy of each will be recorded. Second, dissection and extraction of the sentinel node will be performed, to send it to the frozen section examination. Third, other lymph node could be removed if the surgeon evaluate that it is feasible and necessary. In this group, the false negative rate will be also evaluate.

SUMMARY:
This is an obstervationnal study, to evaluate the good clinical practice of the use of the sentinel node biospy in early stage endometrial cancer. The collaborating centres with the OncoGynecology board of the King Albert II Institute of the Clinique Universitaire Saint-Luc will also particpate to the trial.

Sentinel node biospy is not yet validated for endometrial cancer, even if lots of leading team in the world published very good result and that the first prospectives trials are already published with also excellents results. The investigators decided then to include this practice in their institutional guideslines and also to registred the procedure.

DETAILED DESCRIPTION:
All the sentinel node biopsy procedures for endometrial cancer will be record online via the REDCap tools, securized on a servor in Saint-Luc. Automatic email for the following of the patients and the post operative event will be send regularly for every patient to the physicians who include the patient. Efficacy of the technique, False negative and postive rate, modifications of the adjuvant treatement, long terme evolution and complication wil be evaluate.

ELIGIBILITY:
Inclusion Criteria:

* Endometrial cancer early stage on the pre operative examinations
* Performance status that allow a surgery
* Surgery by laparoscopy or laparotomy

Exclusion Criteria:

* Patient already operated of the hysterectomy who need lymphatic restadification
* Stage IV disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All the patient with early stage endometrial cancer, whith or without indication of complete lymphadenectomy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-08; Primary Completion 2020-08 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Detection rate of the sentinel lymph node biopsy regarding diffrent methods used by the investigators | 5 years
  Each hemi pelvis is count as an unit for the detection rate, but also the detection per patient will be calculated. For a positive detection with the patient as an unit, the detection must be bilateral

SECONDARY OUTCOMES:
Modification of the adjuvant treatement by the information bring by the sentinel node analysis | 5 years
  An evaluation of the modification of the adjuvant treatement by the results of the node sentinel will be performed, in case of it was performed alone and then compared to the guides lines when no information on the nodal status is knowed. It will also be evaluated in cas where a complete lymphadenectomy was performed to evaluate the interest of the ultrastaging on the sentinel node.
Survival outcomes: Disease free survival (DFS) and Overvall survival (OS) will be evaluate. | 5 years
  Influence of the use of the sentinel node only or in addition to the complete lymphadenectomy on the DFS and the OS by comparing with the litterature accorded DFS and OS will be evaluate. Type of reccurence will also be attentively observed, in order to ensure the safety of the sentinel node dissection only. If the technique is reliable, the rate of nodal reccurence after negative sentinel node should be low.
False positive rate of the frozen section analysis | 5 years
  Each negative sentinel node at the frozen section analyse wil also undergo a second analysis after "calssical" preparation of the tissue and alos immunochemestry analysis
False negative rate of the sentinel node, after frosen section analyse and the complete analysis | 5 years
  In the group of patient who underwent a complet lymphadenectomy, a false negative rate will be calculate, with a expected number really low.
Early and late complications of the procedure | 5 years
  Per operative, early and late post operative complication related to the sentinel node procedure will be recorded in the REDCap file, and will be compared to the group of complete lymphadenectomy, with a special focus on lymphatics complications (lymphocyst, lymphoedema,...)

CONTACTS AND LOCATIONS:
Overall Officials: Luyckc Luyckx, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (10):
- Belgium (10):
  - CHU AMbroise Parée, Mons, Hainaut
  - Cliniques de l'Europe, Brussels
  - Cliniques universitaires Saint-Luc, Brussels
  - Clinique St Jean, Brussels
  - Cliniques Saint-Anne - Saint Remi, Brussels
  - Hôpital d'Ixelles, Brussels
  - GHDC, Charleroi
  - Université de Liège, Liège
  - Cliniques Saint-Pierre Ottignies, Ottignies
  - CHWaPi, Tournai